CLINICAL TRIAL: NCT03485768
Title: Therapeutic Effects and Safety of Percutaneous Disc Decompression With Coblation Nucleoplasty in Cervical Vertigo
Brief Title: PDCN for Treatment of Cervical Vertigo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Limin Rong, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDCN-CV
Record Dates: First submitted 2018-02-25; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Cervical Vertigo
Keywords: cervical vertigo; percutaneous disc decompression with coblation nucleoplasty; manual therapy; clinical efficacy; randomized controlled trial
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: This is a prospective, one-center, controlled clinical study with random assignment to PDCN or manual therapy group to explore their effectiveness and safety for the treatment of cervicogenic dizziness. Participants will be randomized and allocated to either PDCN group or manual therapy group with 1:1 ratio and with 35 patients in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutaneous disc decompression with coblation nucleoplasty (Experimental): PDCN will be performed in patients who are allocated to this group by using the COBLATION Perc-DC SpineWand surgical device (ArthroCare System 2000, ArthroCare corporation, Heredia, Costa Rica, USA)
  Interventions: Procedure: percutaneous disc decompression with coblation nucleoplasty
- Manual Therapy (Active Comparator): Participants who are allocated to this group will undergo manual therapy treatments containing two kinds: sustained natural apophyseal glides (SNAGs) plus passive joint mobilisations (PJMs)
  Interventions: Procedure: Manual Therapy (SNAGs plus PJMs)

INTERVENTIONS:
Procedure: percutaneous disc decompression with coblation nucleoplasty — PDCN was performed using the COBLATION Perc-DC SpineWand surgical device (ArthroCare System 2000, ArthroCare corporation, Heredia, Costa Rica, USA) under local anesthesia. The introducer cannula was then pierced into the target intervertebral disc through an anterior lateral approach. The tip of the cannula stylet was aimed for the center of the nucleus in both the coronal and sagittal planes. The stylet was withdrawn from the introducer cannula and replaced with the Perc-DC SpineWand. The wand was advanced until its tip extended approximately 5 mm beyond the tip of the cannula. A short initial coagulation was performed upon wand insertion to ensure correct placement, if stimulation or movement was detected, the wand was repositioned. As the wand was drawn back out through the disc, ablation energy was set to level three and three ablation cycles of 5-12soconds each were performed, rotating the wand tip 180 degree each time to form three consecutive pockets within the disc.
  Other Names: PDCN
  Arms: percutaneous disc decompression with coblation nucleoplasty
Procedure: Manual Therapy (SNAGs plus PJMs) — (1) sustained natural apophyseal glides (SNAGs): Use the methods described in Mulligan BR. Manual therapy "NAGS", "SNAGS", "MWMS" etc. 5th ed. Wellington, New Zealand: Plane View Services; 2004. Three sessions per week and for a total of four to six weeks according to the patients' condition, they were asked to continue the self-SNAG once daily until the last follow-up, and recorded in a diary. (2) passive joint mobilisations (PJMs): Use the methods described in Maitland G. Vertebral manipulation. 6th ed. Oxford: Butterworth Heinemann; 2001. For three repetitions weekly and for a total of four to six weeks according to the patients' condition, then once a day were commenced as a home exercise to be continued until the last follow-up, and recorded in a diary.
  Other Names: SNAGs together with PJMs
  Arms: Manual Therapy

SUMMARY:
This is a prospective, randomized controlled trial in a single center to explore the effectiveness and safety of percutaneous disc decompression with coblation nucleoplasty (PDCN) for the treatment of cervicogenic dizziness.

DETAILED DESCRIPTION:
Vertigo ranks among the most common complaints in medicine and have a considerable personal impact, affecting 15-35% of the general population at some point in their lives. The combination of neck disorders with vertigo or dizziness was formally coined "cervical vertigo" by Ryan and Cope in 1955. The precise incidence of cervical vertigo is controversial but it is estimated that 20-58% of patients who sustain closed-head injuries or whiplash experience late onset symptoms of dizziness, vertigo and disequilibrium. The treatment option of cervical vertigo is versatile and challenging. Surgical intervention is recommended when the patient is a good candidate. Plasma-mediated ablation using the Coblation Spine-Wand device has been used for several years to perform spine disc decompression. However, there is no short and long-term report of percutaneous disc decompression with coblation nucleoplasty (PDCN) for treatment of cervical vertigo, and complications observed with this procedure have not been reported yet. In the retrospective observational study (unpublished data), the investigators found that PDCN was effective for reducing cervicogenic dizziness, a disabling and persistent problem, in the long term. A mean effective rate of 94.6% (70 of the 74 patients) one week after surgery and 90.6% (67 of the 74 patients) at the last follow-up (1 year to 8 years and 3 months). Good to excellent results were attained in 85.1% (63 of the 74 patients) of these patients one week after PDCN and achieved in 75.7% (56 of the 74 patients) at the last follow-up (p<0.0001). Recently, a randomized trial had proven that manual therapy had long-term beneficial effects in the treatment of chronic cervicogenic dizziness. This study aims to conduct a randomized controlled trial to investigate both of its short term and long term effectiveness and safety in prospective fashion comparing with manual therapy. Participants will be randomized and allocated to either PDCN group or manual therapy group with 1:1 ratio. All the patients had recurring symptom of dizziness over three months and conservative treatment applied for at least three weeks and failed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervical vertigo upon characteristic symptoms of dizziness associated with neck stiffness and/or neck pain, which is related to movement or position of cervical spine;
* Subjects with obvious disc degeneration verified to exist at MRI;
* All the patients had recurring symptom of dizziness over three months and conservative treatment applied for at least three weeks and failed;
* Male or female aged between 18 and 80;
* Subjects' consent to participate and had signed the informed consent.

Exclusion Criteria:

* Other causes of vertigo, including those arising from disturbances of the ear, nose, and throat (ENT); benign positional paroxysmal vertigo (BPPV); central nervous system (CNS); and cardiovascular system;
* Predominant radiculopathy cervical, cervical myelopathy or cervical stenosis;
* Inflammatory arthritis, neoplastic diseases, infection, trauma;
* History of previous cervical surgeries or cervical spine surgery during the follow-up period;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of baseline in Dizziness Intensity | Change between Baseline and 1 week- 1 month- 3 months- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  Self-reported dizziness on a 100mm visual analogue scale (VAS)

SECONDARY OUTCOMES:
Dizziness frequency (rated between o (none) and 5 (>once/day)) | Change between Baseline and 1 week- 1 month- 3 months- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  Self-reported dizziness on a scale of 0-10
Change in Dizziness Handicap Index (DHI) Score | Change between Baseline and 1 week- 1 month- 3 months- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  Self-reported measure evaluating perceived handicap secondary to dizziness, the DHI has 25 items with 3 response levels, sub-grouped into three domains: functional, emotional, and physical
Change in Numeric Pain Rating Scale Score-Neck pain | Change between Baseline and 1 week- 1 month- 3 months- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  Self-report score for headache on a scale of 0-10
Change in SF-36 Health Scale Score | Change between Baseline and 1 week- 1 month- 3 months- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  Self-report score for assessing both of physical functioning and bodily pain on a scale of 12 items
Clinical efficacy assessed by 10 point rating scale | 1 week- 1 month- 3 months- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  0=no benefit, 1=minimal benefit, 2=some benefit, 3=a lot of benefit, 4=great benefit, 5=maximal benefit
Clinical efficacy evaluated by modified MacNab evaluation criteria | 1 week- 1 month- 3 months- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  excellent (A)=dizziness and associated symptoms disappeared completely, resumed normal work and life; good (B)= improved significantly, could do former work; acceptable (C)=somewhat improved, could only undertake light work; poor (D)=not improved significantly, further treatment was required. Fitness rate=A+B; Effective rate=A+B+C
Surgical complications | during operation, up to 1 week and 1 month and 3 months and 6 months respectively after intervention
  discitis, neurological complications, vascular injuries, dural Injury, CSF Leakage, recrudescence, and other severe adverse effects
Image findings evaluated by Magnetic Resonance Imaging | Change between Baseline and 1 week- 1 month- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  changes of intervertebral disc signal and herniation
Changes of intervertebral disc height assessed by X ray | Change between Baseline and 1 week- 1 month- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  height of anterior, middle and posterior portion of the targeted disc (disc with intervention)
Changes of cobb angle assessed by X ray | Change between Baseline and 1 week- 1 month- 6 months- 1 year- 2 years- 3 years- 5 years respectively after treatment
  draw a line either parallel to the inferior endplate of C-2 or extending from the anterior tubercle of C-1 to the posterior margin of the spinous process, and another line parallel to the inferior endplate of C-7. Perpendicular lines are then drawn from each of the 2 lines noted above, and the angle subtended between the crossing of the perpendicular lines is the cervical curvature angle

CONTACTS AND LOCATIONS:
Overall Officials: Limin Rong, Ph.D, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neuhauser HK. The epidemiology of dizziness and vertigo. Handb Clin Neurol. 2016;137:67-82. doi: 10.1016/B978-0-444-63437-5.00005-4. PMID 27638063
- [Background] RYAN GM, COPE S. Cervical vertigo. Lancet. 1955 Dec 31;269(6905):1355-8. doi: 10.1016/s0140-6736(55)93159-7. No abstract available. PMID 13279136
- [Background] Wenngren BI, Pettersson K, Lowenhielm G, Hildingsson C. Eye motility and auditory brainstem response dysfunction after whiplash injury. Acta Otolaryngol. 2002 Apr;122(3):276-83. doi: 10.1080/000164802753648150. PMID 12030574
- [Background] Endo K, Ichimaru K, Komagata M, Yamamoto K. Cervical vertigo and dizziness after whiplash injury. Eur Spine J. 2006 Jun;15(6):886-90. doi: 10.1007/s00586-005-0970-y. Epub 2006 Jan 24. PMID 16432749
- [Background] Endo K, Suzuki H, Yamamoto K. Consciously postural sway and cervical vertigo after whiplash injury. Spine (Phila Pa 1976). 2008 Jul 15;33(16):E539-42. doi: 10.1097/BRS.0b013e31817c55fe. PMID 18628694
- [Background] Li Y, Peng B. Pathogenesis, Diagnosis, and Treatment of Cervical Vertigo. Pain Physician. 2015 Jul-Aug;18(4):E583-95. PMID 26218949
- [Background] Cesaroni A, Nardi PV. Plasma disc decompression for contained cervical disc herniation: a randomized, controlled trial. Eur Spine J. 2010 Mar;19(3):477-86. doi: 10.1007/s00586-009-1189-0. Epub 2009 Nov 10. PMID 19902277
- [Background] Masala S, Massari F, Fabiano S, Ursone A, Fiori R, Pastore F, Simonetti G. Nucleoplasty in the treatment of lumbar diskogenic back pain: one year follow-up. Cardiovasc Intervent Radiol. 2007 May-Jun;30(3):426-32. doi: 10.1007/s00270-006-0223-4. PMID 17278033
- [Background] Gerszten PC, Smuck M, Rathmell JP, Simopoulos TT, Bhagia SM, Mocek CK, Crabtree T, Bloch DA; SPINE Study Group. Plasma disc decompression compared with fluoroscopy-guided transforaminal epidural steroid injections for symptomatic contained lumbar disc herniation: a prospective, randomized, controlled trial. J Neurosurg Spine. 2010 Apr;12(4):357-71. doi: 10.3171/2009.10.SPINE09208. PMID 20201654
- [Background] Nikoobakht M, Yekanineajd MS, Pakpour AH, Gerszten PC, Kasch R. Plasma disc decompression compared to physiotherapy for symptomatic contained lumbar disc herniation: A prospective randomized controlled trial. Neurol Neurochir Pol. 2016;50(1):24-30. doi: 10.1016/j.pjnns.2015.11.001. Epub 2015 Nov 28. PMID 26851686
- [Background] Eichen PM, Achilles N, Konig V, Mosges R, Hellmich M, Himpe B, Kirchner R. Nucleoplasty, a minimally invasive procedure for disc decompression: a systematic review and meta-analysis of published clinical studies. Pain Physician. 2014 Mar-Apr;17(2):E149-73. PMID 24658486
- [Background] Reid SA, Callister R, Snodgrass SJ, Katekar MG, Rivett DA. Manual therapy for cervicogenic dizziness: Long-term outcomes of a randomised trial. Man Ther. 2015 Feb;20(1):148-56. doi: 10.1016/j.math.2014.08.003. Epub 2014 Aug 27. PMID 25220110